CLINICAL TRIAL: NCT06072950
Title: Opioid Use and Predicting Factors at the Emergency Department
Acronym: VRxOPUS-1
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 113728
Record Dates: First submitted 2023-09-18; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Pain; Pain, Acute
Keywords: Emergency Department; Pain at rest; Opioid use
MeSH Terms: conditions — Pain; Acute Pain; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with NRS pain at rest being 4 or higher: Patient with NRS pain at rest being 4 or higher, primarily treated by emergency physician, internist, or surgeon. All patients receive usual care, no interventions are administered.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Usual care — Patients received usual care

SUMMARY:
Background: Increasing opioid misuse is a worldwide problem. About 10% of opioid misusers are primarily exposed to opioids at the Emergency Department (ED). This study was conducted to determine the feasibility for a clinical trial investigating the effect of Virtual Reality therapy on opioid consumption at the ED.

Methods: Adult patients were included when primarily seen by the Emergency Physician and presenting with a NRS pain score ≥4. Main objective was to identify the target population and evaluate outcome measures to sustain a trial incorporating the Oral Morphine Equivalent (OME) at the ED as the primary endpoint. Primary outcome was mean OME administered at the ED. Secondary outcomes included NRS pain scores, main symptoms and type of analgesics administered at the ED.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥16 years admitted to ED and identified by an Emergency Physician (EP)
* NRS pain score ≥4
* Patient is willing and able to comply with the study protocol

Exclusion Criteria:

* Patients initially treated by another physician than the EP.
* EMV < 14
* History of dementia, seizures
* Severe hearing/visual impairment not corrected
* Headwounds or damaged skin with which comfortable and hygienic use is not possible.
* Presentation to ED because of chronic pain (≥3 months) exacerbation
* Chronic opioids use (≥3 months)

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We aim to include all patients ≥16 years, who are admitted to the ED of the Radboudumc and primarily seen by an ED physician.
Sampling Method: Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Opioid use | throughout study participation, up to 8 hours
  Opioids use of patients during their stay at Emergency Department (yes/no)

SECONDARY OUTCOMES:
Oral morphine equivalent | throughout study participation, up to 8 hours
  Doses of opioids received by a patient during their stay at the ED converted to Oral morphine equivalent (OME)
Administered analgesics | throughout study participation, up to 8 hours
  Type and dose of all administered analgesics at Emergency Department.
Pain acceptability | Asked at moment of admittance and at discharge, up to 6 hours after inclusion
  Patient opinion on acceptability of their pain at rest upon admittance and discharge
Reason why patients finds pain acceptable | Assessed upon admittance
  Open question
Patients desire for analgesics | Asked at moment of admittance and at discharge, up to 6 hours after inclusion
  yes/no question whether patient desires analgesics
Patients openness to VR | Assessed upon admittance
  yes/no question to explore patients willingeness to use VR in their situation
Numaric rating score pain scores at rest | Every 30 minutes until discharge of patient
  Including whether this is pre/post analgesics
Numaric rating score anxiety scores | Every 30 minutes until discharge of patient
  NRS anxiety scores
Satisfaction with pain management | Asked at moment of discharge, up to 6 hours after inclusion
  On a numaric rating scale
Nurse opinion on patient adequacy of pain reporting | Assessed upon admittance
  Categorical question: understating - adequate - exaggerating
Duration of ED visit | throughout study participation, up to 8 hours
  Duration of ED visit
Analgesics prescriptions | throughout study participation, up to 8 hours
  When patient is discharged home prescribed analgesics are registered.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon reasonable request.